CLINICAL TRIAL: NCT01471106
Title: Phase II Short-term Adjuvant Therapy and Biomarker Studies With Targeted Agents in Women With Estrogen Receptor Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0794; NCI-2012-00037 (Registry Identifier: NCI CTRP); KG09 1020 (Other: Susan G. Komen Breast Cancer Foundation)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Estrogen Receptor Negative Breast Cancer; Biomarker studies; Ki-67; Dasatinib; BMS-354825; Sprycel
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Dasatinib 40 mg (Experimental): Dasatinib 40 mg by mouth once a day for 3 months (+/- 7 days), At the end of the 3 months (+/- 7 days) participants undergo a repeat FNA and blood collection for the same marker analyses.
  Interventions: Drug: Dasatinib
- Group 3: No Dasatinib (No Intervention): No treatment control group. At the end of the 3 months (+/- 7 days) participants undergo a repeat FNA and blood collection for the same marker analyses.
- Group 2: Dasatinib 80 mg (Experimental): Dasatinib 80 mg by mouth once a day for 3 months (+/- 7 days). At the end of the 3 months (+/- 7 days) participants undergo a repeat FNA and blood collection for the same marker analyses.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Group 1: 40 mg by mouth once a day.
  Group 2: 80 mg by mouth once a day.
  Other Names: BMS-354825; Sprycel
  Arms: Group 1: Dasatinib 40 mg; Group 2: Dasatinib 80 mg

SUMMARY:
The goal of this clinical research study is to learn if dasatinib can help prevent breast cancer from developing in the unaffected breast.

Dasatinib is designed to decrease the activity of one or more proteins that are responsible for the uncontrolled growth of tumor cells.

This is an investigational study. Dasatinib is FDA approved and commercially available for the treatment of leukemia. Its use in breast cancer patients in investigational.

Up to 66 patients will take part in this multicenter study. Up to 60 will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 3 study groups:

* If you are in Group 1, you will take dasatinib 40mg once a day by mouth with water.
* If you are in Group 2, you will take dasatinib 80mg once a day by mouth with water.
* If you are in Group 3, you will not receive dasatinib.

You will be given a study drug diary to complete. In the diary, you will record when you take the study drug.

Study Visits:

At Month 1:

* You will be called by a nurse and asked about any drugs you are taking and side effects you may be having.
* You will be asked about any drugs you may be taking and side effects you may be having.
* Your drug diary will be reviewed.

At Month 2 you will be called by a nurse and asked about any drugs you are taking and side effects you may be having. You will also be asked to review your drug diary. This call will take about 20 minutes

At Month 3 (or if you leave the study early):

* You will have a fine needle aspirate (FNA) of the breast for biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.
* Blood (about 2-3 tablespoons) will be drawn for biomarker testing.
* You will be asked about any drugs you may be taking and side effects you may be having.
* Your drug diary will be reviewed.

Length of Study:

You may remain on study for up to 3 months. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of ER negative breast carcinoma (defined as less than 10%), stage I, II, or III
2. Completed all adjuvant therapy including (if indicated) endocrine, trastuzumab, radiation therapy
3. At least 18 years of age.
4. Female: A female is eligible to enter and participate in the study if she is of: a. Non-childbearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation, hysterectomy alone, hysterectomy and bilateral salpingo-oophorectomy, bilateral salpingo-oophorectomy alone or women who are post-menopausal); or b. Childbearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility. This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate), has a negative serum pregnancy test at screening, and agrees to one of the following where considered acceptable to the local IRB/IEC: • Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm).
5. (Continued from above) • Abstinence from sexual intercourse from 2 weeks prior to administration of the investigational product, throughout the active study treatment period. • Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject. • Any intrauterine device (IUD). • Barrier methods including diaphragm or condom with a spermicide.
6. Able to swallow and retain oral medication.
7. ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2.
8. Provided written informed consent.
9. Adequate bone marrow function: Hemoglobin >/= 9 gm/dL. • Absolute granulocyte count >/= 1,500/mm^3 (1.5 x 10^9/L). • Platelets >/= 75,000/mm^3 (100 x 10^9/L).
10. Serum creatinine < 1.4 mg/dL or calculated creatinine clearance (CrCl) >/= 30 mL/min
11. Total bilirubin </= 1.5 times the upper limit of the reference range
12. Aspartate and alanine transaminase (AST or ALT) </= 2 times the upper limit of the reference range.
13. Patients must have a baseline ECG with QTcF within the normal range within 28 days prior to registration.
14. Normal mammogram of unaffected breast within 12 months prior to study entry.

Exclusion Criteria:

1. Unwillingness to undergo RPFNA.
2. Contraindication to RPFNA including breast implant(s), bilateral radiation, anticoagulation (excluding those on 81mg aspirin).
3. Concurrent medical condition that would increase drug toxicity: Pleural or pericardial effusion, coagulation or platelet function disorder, ongoing or recent (less than 3 months gastrointestinal bleeding)
4. Uncontrolled angina, congestive heart failure, MI (within last 6 months), congenital long QT syndrome, history of clinically significant ventricular arrhythmia, prolonged QTcF interval on pre-entry EKG (greater than normal range)
5. Hypokalemia or hypomagnesemia if it cannot be corrected
6. Is a pregnant or lactating female.
7. Has evidence of recurrent or metastatic (Stage IV) breast cancer.
8. Is considered medically unfit for the study by the investigator as a result of the medical interview, physical exam, or screening investigations.
9. Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to dasatinib
10. Has received treatment with any investigational drug in the previous 4 weeks.
11. Has received chemotherapy, immunotherapy, biologic therapy or endocrine therapy within the past 12 weeks.
12. Is currently receiving oral steroid treatment (inhaled steroids are permitted)
13. Oral estrogen, progesterone, testosterone therapy within last 3 months.
14. Concomitant Medications: Drugs that are considered category D (Consider therapy modification) and X (Avoid combination) using the Lexicomp database are prohibited. Concomitant drugs that fall into categories A (No known interaction), B (no action needed) and C (monitor therapy) are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 patients were enrolled by 08/13/2018, of which were 24 randomized, 6 in No Treatment/Control, 12 in Dasatinib 40 mg, and 6 in Dasatinib 80 mg.
Groups:
- Group 1: Dasatinib 40 mg: Dasatinib 40 mg by mouth once a day for 3 months (+/- 7 days), At the end of the 3 months (+/- 7 days) participants undergo a repeat FNA and blood collection for the same marker analyses.
  Dasatinib: Group 1: 40 mg by mouth once a day.
  Dasatinib Group 2: 80 mg by mouth once a day.
- Group 2: Dasatinib 80 mg: Dasatinib 80 mg by mouth once a day for 3 months (+/- 7 days). At the end of the 3 months (+/- 7 days) participants undergo a repeat FNA and blood collection for the same marker analyses.
  Dasatinib: Group 1: 40 mg by mouth once a day.
  Dasatinib Group 2: 80 mg by mouth once a day.
Period: Overall Study
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
Started | 12 | 6 | 6
Completed | 12 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib | Total
Number analyzed (Participants) | 12 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 6 | 23
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Median (Full Range); unit: Years] | 62.4 [46.1 to 74.4] | 50.8 [30.7 to 69.6] | 54 [40.6 to 63.2] | 56.8 [30.7 to 74.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 6 | 24
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 9 | 5 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 10 | 4 | 4 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki-67 in Breast Tissue of High-Risk Women
Description: Change in Ki-67 measured in baseline and month 3 using contralateral breast Fine Needle Aspiration (FNA) samples. Samples evaluated by immunohistochemistry (IHC). Baseline and follow up Ki-67 values presented in percentage (%) of cell positive, change reflects difference in percentage. Ki-67 is measured as a continuous variable and a one-way ANOVA followed by Dunnett's multiple comparison test comparing the change of Ki-67 of each of the three treated groups with control.
Time Frame: up to 3 months
Population: FNA yield for matched pre-and-post treatment FNA samples was technically insufficient for Ki-67 immunohistochemitry analysis
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: To Evaluate Dasatinib Induced Modulation of Biomarker in the Serum Including Insulin Like Growth Factor (IGF) Pathway
Description: Evaluation of serum utilizing ELISA kits for IGFBP1
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
Number analyzed (Participants) | 12 | 6 | 6
pg/ml
  Pre-treatment | 6683 (4086.6) | 2320.9 (797.1) | 6524 (3900.3)
  Post-treatment | 8508.5 (7992.3) | 4270.6 (4405.3) | 7270.1 (4715.4)

3. Secondary Outcome: To Evaluate Dasatinib Induced Modulation of Biomarker in the Serum Including Insulin Like Growth Factor (IGF) Pathway
Description: Evaluation of serum utilizing ELISA kits for IGF1
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
Number analyzed (Participants) | 12 | 6 | 6
ng/ml
  Pre-treatment | 71.8 (35.6) | 79.8 (22.3) | 95.2 (25.7)
  Post-treatment | 70.3 (41) | 68.2 (24.4) | 95.3 (27.7)

4. Secondary Outcome: To Evaluate Dasatinib Induced Modulation of Biomarker in the Serum Including Insulin Like Growth Factor (IGF) Pathway
Description: Evaluation of serum utilizing ELISA kits for IGFBP3
Time Frame: up to 3 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
Number analyzed (Participants) | 12 | 6 | 6
ng/ml
  pretreatment | 2041 (411.1) | 1999 (136.7) | 2279.9 (394.5)
  Post-treatment | 2027.6 (348.9) | 2048.4 (220.7) | 2080.2 (514.4)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Group 1: Dasatinib 40 mg | Group 2: Dasatinib 80 mg | Group 3: No Dasatinib
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 11/12 | 5/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Dasatinib 40 mg (N=12) | Group 2: Dasatinib 80 mg (N=6) | Group 3: No Dasatinib (N=6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - (Other), specify (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 2 (2) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - (Other), specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Specify (Other) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - (Other), specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT01471106/Prot_SAP_000.pdf